CLINICAL TRIAL: NCT00345891
Title: Quite Smoking Program for Lung Cancer Patients' Families
Brief Title: Quit Smoking Program for Lung Cancer Patients' Families (The Family Ties Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008930; U01CA092622 (NIH)
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2010-05

CONDITIONS: Smoking Cessation
Keywords: Lung neoplasms; Family; Stress
MeSH Terms: conditions — Smoking Cessation; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Coping-focused counseling telephone calls

SUMMARY:
The purpose of this study is to evaluate the impact of delivering a coping-focused intervention as an adjunct to a self-help program to promote smoking cessation among relatives of lung cancer patients.

DETAILED DESCRIPTION:
Despite the fact that lung cancer is attributed almost entirely to cigarette smoking and smoking cessation substantially decreases the risk for lung cancer, many smokers are not significantly motivated to quit smoking. A loved one's diagnosis of terminal lung cancer diagnosis presents a time when relatives who smoke are in need of and may be especially receptive to smoking cessation interventions.

The overarching aim of the study is to evaluate in a randomized trial the impact of delivering a coping-focused intervention as an adjunct to a state-of-the-science self-help program to promote smoking cessation among relatives of lung cancer patients. The specific aims are as follows:

1. To evaluate the impact of a coping-focused self-help intervention on relatives' rates of abstinence from cigarettes at 2 weeks, 6- and 12-months post-treatment follow-ups.
2. To evaluate whether any observed intervention effect on abstinence rates is mediated by improvements in relative's cognitive appraisals specifically self-efficacy, and perceived control over health outcomes, adaptive coping responses, and decreases in stress and depression
3. To evaluate the cost-effectiveness of the standard self-help and coping-focused interventions.

Patient diagnosed with lung cancer will be contacted and asked to enumerate their relatives (i.e., immediate family, extended family, spouses, and anyone perceived as family) and asked the smoking status of each of these relatives. Patients will then be asked for permission to send their relatives who smoke a letter that describes the study and provides a telephone number to call to decline participation. Patients who are current smokers may receive materials to help them stop smoking.

The relatives who do not call to decline participation will be contacted by the survey company to ask them to participate in a telephone survey. If eligible and willing, verbal consent will be obtained from relatives who smoke to complete the 20-30 minute baseline survey. During the telephone contact, relatives will have the opportunity to decline to complete the survey and to be further involved in the research study.

The first relative in a family who participates will be randomized to one of two intervention arms: Standard self-help (N=240) or Coping-focused self-help (N=240). Once randomized, patients will receive the following intervention:

STANDARD SELF-HELP: Relatives who smoke will receive a letter from the clinic where their family member receives care to encourage smoking cessation and to introduce the study. A tailored booklet that encourages the relative to quit smoking will introduce a self-help quit kit (e.g., written cessation booklet, audio relaxation tape, over-the-counter nicotine patches, if applicable).

COPING-FOCUSED SELF-HELP: Participants in this arm will receive a letter from the clinic where their family member receives care (i.e. TOP, MTOP, or MTOC), tailored booklet and self-help quit kit. In addition, these relatives will receive a total of six counseling phone calls that will be delivered in tandem with the tailored materials. Optimally these phone calls will be scheduled once a week for a total of six weeks in order to retain participation and to encourage practice and use of skills covered during the phone calls. All calls must be completed with a 12-week period. Each intervention component will emphasize: the salience of the patient's diagnosis as a prompt for smoking cessation or to maintain abstinence and the importance of coping in ways that promote successful smoking cessation.

All family members will be surveyed at baseline, 2 weeks, 6 months and 12- months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria-Patients:
* Diagnosis of lung cancer
* Ages 18 or older
* Able to consent

Inclusion Criteria-Family Members:

* Patient has given consent to contact the family member
* Ages 18 or older
* Speaks and reads English
* Cognitively able to give consent to participate
* Has access to a telephone
* Smoked at least 100 cigarettes in his/her life
* Smoked any cigarettes in the prior 7 days at screening

Exclusion Criteria:

* Patients or family members who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
7-day point-prevalence abstinence at 2 weeks and 6 month follow-up

SECONDARY OUTCOMES:
7-day point-prevalence abstinence at the 12-month follow-up and prolonged abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Bastian, MD, MPH, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - H. Lee Moffitt Cancer Center & Research Institute Thoracic Oncology Program, Tampa, Florida
  - UNC Chapel Hill Multidisciplinary Thoracic Oncology Program, Chapel Hill, North Carolina
  - Durham VAMC Medical Thoracic Oncology Clinic, Durham, North Carolina
  - Duke University Medical Center Thoracic Oncology Program, Durham, North Carolina

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Bastian LA, Fish LJ, Peterson BL, Biddle AK, Garst J, Lyna P, Molner S, Bepler G, Kelley M, Keefe FJ, McBride CM. Assessment of the impact of adjunctive proactive telephone counseling to promote smoking cessation among lung cancer patients' social networks. Am J Health Promot. 2013 Jan-Feb;27(3):181-90. doi: 10.4278/ajhp.101122-QUAN-387. PMID 23286595